CLINICAL TRIAL: NCT04115956
Title: An Open-Label, Phase 1/2 Study of Melflufen and Dexamethasone for Patients With AL Amyloidosis Following at Least One Prior Line of Therapy
Brief Title: A Clinical Study of Melphalan Flufenamide (Melflufen) and Dexamethasone for Patients With Immunoglobulin Light Chain (AL) Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study following an FDA request of a partial clinical hold.
Sponsor: Oncopeptides AB (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP201
Record Dates: First submitted 2019-08-29; First posted 2019-10-04 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-02

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — melflufen; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Melflufen + Dexamethasone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Melflufen and dexamethasone in combination (Experimental): Intravenous infusion of melflufen Day 1 of 28 day cycles, in combination of dexamethasone on Days 1 and 2 of each 28-day cycle.
  Interventions: Drug: Melphalan-Flufenamide (Melflufen); Drug: Dexamethasone

INTERVENTIONS:
Drug: Melphalan-Flufenamide (Melflufen) — Treatment consist of i.v. melflufen on Day 1 of each 28-day cycle.
Drug: Dexamethasone — Dexamethasone 40 mg (20 mg at investigator's discretion) administered on Days 1 and 2 of each 28-day cycle.
  Other Names: Dexamethason JENAPHARM

SUMMARY:
This is a phase 1/2 open label study of melphalan flufenamide (melflufen) in combination with dexamethasone for participants with Al amyloidosis following at least one prior line of therapy. Melflufen will be administered on Day 1 of each 28-day cycle in combination with dexamethasone on days 1 and 2.

In both phases, treatment of each individual participant will continue for up to 8 cycles or until any stopping events occur.

Approximately 46 participants will be enrolled.

The study was intended to be a Phase 1/2 trial but was early terminated and never moved forward to Phase 2.

DETAILED DESCRIPTION:
This is a clinical trial of melphalan flufenamide (melflufen), a peptide-conjugated alkylator which belongs to an novel class of drugs called peptidase-enhanced compounds, and targets the transformation process of tumor cells with a unique mechanism of action, as potential treatment option of AL amyloidosis.

AL amyloidosis is a rare progressive disease caused by proteotoxic light chain protein produced by small plasma cell clone. This plasma cell dyscrasia is characterized by monoclonal plasma cell's excessive production of monoclonal immunoglobulin light-chains that tends to misfold and subsequently deposit as amyloid fibrils in visceral organs. The plasma cell dyscrasia in AL amyloidosis is similar to that in multiple myeloma (MM) and therapies that are effective in MM are often used to treat AL amyloidosis.

Melphalan flufenamide is currently been evaluated in several ongoing clinical trials in patients with multiple myeloma, with observed efficacy. There are currently no therapies approved for treatment of AL amyloidosis and based on the efficacy of melphalan flufenamide and the demonstrated efficacy of melphalan (and other alkylators), it is anticipated that patients with AL amyloidosis may receive benefit from treatment with melphalan flufenamide.

This study consist of a screening period (up to 28 days), a treatment period (up to 8 cycles) and a follow-up period (up to 24 months).

Phase 1: Approximately 8-30 participants will be screened to achieve 7-23 enrolled participants.

Phase 2: Approximately 30 participants will be screened to achieve 23 enrolled participants.

The study was intended to be a Phase 1/2 trial but was early terminated and study never moved forward to Phase 2.

ELIGIBILITY:
Inclusion Criteria: (For full list of inclusion criteria, see study protocol)

* Male or female, age 18 years or older at the time of signing the informed consent
* Proven histochemical diagnosis of AL amyloidosis based on tissue specimens with Congo red staining
* At least one prior line of therapy, defined as either one non-transplant regimen, one ASCT (autologous stem cell transplantation), or one regimen of induction therapy followed by a single ASCT. No more that 4 cycles of melphalan containing chemotherapy is allowed.
* Measurable hematologic disease
* Objectively measurable organ amyloid involvement
* ECOG performance status ≤ 2 (ECOG = Eastern cooperative oncology group)
* Women of child bearing potential must have a negative serum or urine pregnancy test
* Less than 30% plasma cells in bone marrow aspirate or biopsy
* Acceptable laboratory results met (absolute neutrophil count (ANC), platelet count, hemoglobin, total bilirubin,alkaline phosphatase, AST (aspartate aminotransferase) and ALT (alanine aminotransferase), renal function)
* Male participant agrees to use contraception during treatment and 90 days after last dose of melflufen

Exclusion Criteria: (For full list of exclusion criteria, see study protocol)

* Amyloidosis due to known mutations of the transthyretin gene or presence of another non-AL amyloidosis
* Evidence of gastro-intestinal bleeding
* Cardiac risk stage 3
* Low platelets value with evidence of mucosal or internal bleeding
* Medical documented cardiac syncope, NYHA Class 3 or 4 congestive heart failure, myocardial infarction, unstable angina pectoris, clinically significant ventricular arrhythmias (NYHA=New York Heart Association Functional Classification)
* Clinically significant finding on 24 h Holter recording
* Severe orthostatic hypotension
* Clinically significant factor X deficiency
* Clinically significant autonomic disease
* Any medical condition that would impose excessive risk to the patient
* Serious psychiatric illness, active alcoholism or drug addiction that may hinder or confuse compliance
* Known HIV or active hepatitis B or C viral infections
* Previous cytotoxic therapies, including cytotoxic investigational agents within 3 weeks prior to start of study treatment. Monoclonal antibodies within 4 weeks. Concomitant immunotherapy, investigational therapy and anticoagulation therapy are not permitted
* Prior autologous or allogenic stem cell transplant within 12 weeks of initiation of therapy
* Prior allogeneic stem cell transplant with active graft-host-disease
* Prior major surgical procedure or radiation therapy within 4 weeks of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
The primary objective in Phase 1 is to explore safety and tolerability of melflufen | During phase 1 for up to 8 cycles of treatment of 28 days each (approx. up to 8 months)
  Endpoints:
  * Frequency and grade of Adverse Events. The maximum grade for each type of AE will be recorded for each participant and frequency tables will be presented and reviewed to determine patterns
  * Laboratory values (laboratory abnormalities) for hematology, coagulation, blood chemistry, urinalysis
The primary objective in Phase 1 is to identify recommended Phase 2 dose (RP2D) | During phase 1 for up to 8 cycles of 28 days each (approx. up to 8 months)
  Endpoint: Dose-Limiting Toxicity (DLT) during Cycle 1 up to maximum dose of melflufen of 40 mg. A DLT event is defined as thrombocytopenia, neutropenia, non-hematologic toxicity and/or inability to receive Cycle 2 Day 1 dose within 14 days from planned Cycle 2 Day 2 due to continued melflufen-related toxicity from Cycle 1.
The primary endpoint in Phase 2 is to evaluate the hematologic overall response rate (ORR) after 4 cycles at the RP2D determined in Phase 1 | During phase 2 after 4 cycles of treatment ( approx. 4 months)
  The proportion of participants who achieve a hematologic Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR)

SECONDARY OUTCOMES:
To assess pharmacokinetic profile of melflufen in this patient population | At Cycle 1 Day 1 and Cycle 2 Day 1 at time points 5-10 minutes, 1-2 hours and 3-8 hours after end of infusion. Each cycle length is 28 days.
  Melphalan plasma concentration post melflufen administration at 3 time points
To assess best hematologic response | Throughout the study treatment of up to 8 cycles of 28 days each (approx. 8 months) per patient
  Proportion of patients with each outcome (Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR) or Progressive Disease (PD))
To assess the duration of hematologic response | Throughout the study treatment period of up to 8 cycles of 28 days each (approx 8 months) per patient
  Median time (Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR) or Progressive Disease (PD))
To assess the proportion of organ system responses | Throughout the study treatment period of up to 8 cycles of 28 days each (approx 8 months) per patient
  Proportion of participants with kidney, cardiac or liver response, respectively
To assess duration of organ system responses | Throughout the study treatment period of up to 8 cycles (approx 8 months) per patient
  Duration of organ responses separately for each organ
To assess hematologic ORR (overall response rate) | During phase 1 for up to 8 cycles of treatment of 28 days each (approx. up to 8 months)
  Proportion of participants who achieve a hematologic CR, VGPR or PR
To assess time to next AL amyloidosis treatment | Throughout the study, covering up to 8 cycles (approx. 8 months) of treatment and 24 months of follow up
  Time to next AL amyloidosis treatment
To assess Overall Survival (OS) | Throughout the study, covering up to 8 cycles (approx. 8 months) of treatment and up to 24 months of follow up
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Palladini, MD, Principal Investigator — University Hospital San Matteo in Pavia
Locations (9):
- Boston University Medical Center, Boston, Massachusetts, United States
- Fakultní Nemocnice Ostrava, Ostrava - Poruba, Czechia
- Centre Hospitalier Universitaire de Limoges, Limoges, France
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Alexandra General Hospital of Athens, Athens, Greece
- Hadassah University Hospital Ein Kerem, Jerusalem, Israel
- Oslo University Hospital - Rikshospitalet, Oslo, Norway
- Hospital Clinic de Barcelona, Barcelona, Spain
- University College London Hospitals NHS Foundation Trust, London, United Kingdom